CLINICAL TRIAL: NCT05802433
Title: Effects of VDR rs7311856, GC rs2282679 and CYP2R1 rs2060793 Variants on Vitamin D Status: A Randomised Control Trial
Brief Title: The Genetic Effects on Vitamin D Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Mary's University, Twickenham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SMU_ETHICS_2022-23_004
Record Dates: First submitted 2022-09-14; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Participants are grouped based on their genetic risk of vitamin D deficiency, all participants are given 10µg vitamin D supplements for 90 days
Who Masked: Participant
Masking Description: Participants are not informed of their genetic variations until completion of the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Low risk genotype) (Experimental): Participants with no genetic variation in their VDR, GC and CYP2R1 genes that would increase their risk of vitamin D deficiency. Participants will be given 10µg vitamin D supplements for 90 days. This group is a control against the medium and high-risk intervention groups.
  Interventions: Dietary Supplement: Vitamin D3 supplement
- Intervention (Medium risk genotype) (Experimental): Participants with genetic variation in their VDR, GC and CYP2R1 genes that moderately increase their risk of vitamin D deficiency. Participants will be given 10µg vitamin D supplements for 90 days. This group will be compared against the low-risk control group to determine the effect of genetic variations on vitamin D status.
  Interventions: Dietary Supplement: Vitamin D3 supplement
- Intervention (High risk genotype) (Experimental): Participants with genetic variation in their VDR, GC and CYP2R1 genes that increase their risk of vitamin D deficiency. Participants will be given 10µg vitamin D supplements for 90 days. This group will be compared against the low-risk control group to determine the effect of genetic variations on vitamin D status.
  Interventions: Dietary Supplement: Vitamin D3 supplement

INTERVENTIONS:
Dietary Supplement: Vitamin D3 supplement — 10µg vitamin D3 supplement per day for 90 days

SUMMARY:
Vitamin D is essential for skeletal growth and bone health, deficiency causes rickets and osteomalacia. In the UK 29% of adults have vitamin D deficiency. It is recommended all adults take 10µg vitamin D supplement daily. Genetic variations could alter vitamin D status by affecting vitamin D metabolism. Systematic reviews found variations in VDR, GC and CYP2R1 genes are associated with vitamin D deficiency. This study aims to assess the effects between vitamin D supplementation and variations in VDR, GC and CYP2R1 genes on vitamin D status.

DETAILED DESCRIPTION:
The study design is a quantitative, randomised control trial measuring vitamin D concentrations in blood serum. All participants will be given the recommended 10µg daily dose of vitamin D supplementation. Participants will be grouped based on their genotype for each gene, as either low, medium or high-risk genotypes. The low-risk group will act as a control and the medium and high-risk groups will act as the intervention groups.

Participants will attend St Mary's University's applied science laboratory twice. During their first visit participants will provide a 2ml capillary blood sample. Blood samples are collected using lancets to prick participants' ear lobes. The serum is extracted from the blood samples, serum is stored at -80c until analysis. Participants will be given 90 10µg vitamin D supplements and instructed to take one per day for 90 days. Participants will also be instructed to not make any major changes to their habitual diet. During the second visit participants will provide 1 ml of saliva sample into the Collection Pot and a second 2ml sample of blood. Serum samples will be analysed for vitamin D concentrations using 25(OH) Vitamin D ELISA kit. DNA will be extracted from the saliva samples using PSP SalivaGene DNA Kit following the manufacturer's protocol. DNA will be genotyped for variations in the VDR, GC and CYP2R1 genes. Data will be assessed to determine if variations in these genes influenced the effectiveness of vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* female and male
* 18-65 years
* completion of physical activity readiness questionnaire (PAR-Q).

Exclusion Criteria:

* Below 18 years
* above 65 years
* individuals taking medications that could interact with vitamin D status
* Individuals regularly taking daily Vitamin D supplementation during the 3 months before the intervention start date
* major dietary changes in vitamin D intake during the intervention period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-08-25 (Estimated); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
vitamin D concentration | 90 days
  Effect between genetic variations and vitamin D concentration

CONTACTS AND LOCATIONS:
Overall Officials: Yiannis Mavrommatis, Principal Investigator — St. Mary's University, Twickenham
Locations (1):
- St Mary's University Twickenham, London, Lobdon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krasniqi E, Boshnjaku A, Wagner KH, Wessner B. Association between Polymorphisms in Vitamin D Pathway-Related Genes, Vitamin D Status, Muscle Mass and Function: A Systematic Review. Nutrients. 2021 Sep 4;13(9):3109. doi: 10.3390/nu13093109. PMID 34578986
- [Background] National Health Service (NHS) (2020) Vitamin D. Available at: https://www.nhs.uk/conditions/vitamins-and-minerals/vitamin-d/
- [Background] National Institute for Health and Care Excellence (NICE) (2017) Vitamin D: supplement use in specific population groups. Available at: https://www.nice.org.uk/guidance/ph56/
- [Background] Public Health England (PHE) (2019) National Diet and Nutrition Survey: Years 1 to 9 of the Rolling Programme (2008/2009 - 2016/2017): Time trend and income analyses. Available at: https://assets.publishing.service.gov.uk/
- [Background] Sepulveda-Villegas M, Elizondo-Montemayor L, Trevino V. Identification and analysis of 35 genes associated with vitamin D deficiency: A systematic review to identify genetic variants. J Steroid Biochem Mol Biol. 2020 Feb;196:105516. doi: 10.1016/j.jsbmb.2019.105516. Epub 2019 Oct 31. PMID 31678109